CLINICAL TRIAL: NCT03939455
Title: Mobile Augmented Screening Tool to Increase Adolescent HIV Testing and Linkage to Care
Acronym: MAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Moile Augmented Screening
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: HIV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants will complete a brief tablet-based intervention, which includes watching a 5 minute educational video on the importance of HIV testing, and respond via tablet computer to the offer of an HIV test.
  Interventions: Other: Mobile Augmented Screening tool
- Treatment as usual (No Intervention): Participants will be offered an HIV test by hospital staff, and will respond face-to-face.

INTERVENTIONS:
Other: Mobile Augmented Screening tool — Tablet-based intervention
  Arms: Experimental

SUMMARY:
Because adolescents and young adults face markedly increased HIV risk yet frequently do not test, we propose to complete the Mobile Augmented Screening (MAS) tool designed to increase HIV testing, and to facilitate linkage to care and ongoing prevention education. This tool will help clinicians address undiagnosed youth HIV, and enable young patients to receive much needed treatment and avoid unknowingly transmitting infection. Our product is designed to help existing program staff reach an increased number of clients; and to improve public health by encouraging reluctant young patients to accept important HIV testing and care they may otherwise decline.

DETAILED DESCRIPTION:
Our randomized trial will evaluate HIV test rates among participants who complete a tablet-based intervention, the Mobile Augmented Screening tool (MAS), compared to participants in a treatment as usual (TAU) condition.

Research staff will approach 350 emergency department (ED) patients aged 13 - 24 years. Participants will be randomized into the intervention or TAU condition. Participants will be randomized in a 1:1 ratio to the intervention or TAU condition, stratified by patient age (13-17 and 18-24). Within each of these age strata, permuted blocks randomization with varying block sizes will be employed to ensure balance and concealment of allocations prior to randomization.

Participants who are randomized into the intervention condition will watch a 5-minute video on a tablet computer, and the tablet will ask intervention participants if they would like an HIV test. Possible responses will be "Yes" or "No". Participants who are randomized into TAU will be offered HIV tests by research staff. All participants in both conditions who agree to HIV testing will be tested by hospital staff in the location where they are receiving treatment. All participants who test will receive their results in person from ED staff before discharge.

The primary trial outcome will be percentages of patients, by treatment group, who test for HIV.

ELIGIBILITY:
Inclusion Criteria:

Emergency Department patients aged 13 - 24 years will be eligible for the study if they are:

* awake
* able to provide consent as determined by ED staff
* understand written and spoken English
* not intoxicated
* not known to be HIV positive
* not a prisoner
* have not already agreed to test for HIV during their current ED visit (this will include patients who decline HIV testing offered by hospital staff and patients who are not yet offered HIV testing; potential differences in test rates among participants who decline vs. those who have not previously been offered an HIV test will be explored as a secondary outcome)

Exclusion Criteria:

Exclusion criteria include patients who are prisoners, patients who are asleep/unconscious, unable to provide consent as determined by ED staff, do not understand written and spoken English, are intoxicated, are known to be HIV positive, have already agreed to an HIV test during their current ED visit, have been categorized by ED staff as altered mental status or are presenting to the ED for a psychiatric problem. Additionally, the proposed research will exclude patients if medical records indicate hospital staff have categorized the patient as most urgently in need of medical care.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 295 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
HIV testing | Day of study participation.
  The main outcome is participant HIV testing. We will measure whether the participant accepts an HIV test when offered. Possible outcomes are Yes or No.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

DOCUMENTS (2):
  • Informed Consent Form: Child Assent (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT03939455/ICF_000.pdf
  • Informed Consent Form: Adult Consent (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT03939455/ICF_001.pdf